CLINICAL TRIAL: NCT00340457
Title: Case-Control Study of Renal Cell Cancer Among Caucasians and African Americans in the United States
Brief Title: Case-Control Study of Renal Cell Cancer Among Caucasions and African Americans in the United States
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902051; 02-C-N051; NCT00546338 (obsolete NCT alias); NCT01338220 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma
Keywords: Case-Control Study; Renal Cell Carcinoma; Kidney Cancer; Diet; Occupation
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases: African American patients with renal cancer from two geographic areas of the US
- Controls: African American participants without renal cancer from two geographic areas of the US

SUMMARY:
Incidence rates of renal cell cancer have increased rapidly in the U.S. and other countries. In particular, rates among African Americans have risen more sharply than any other cancer site. We propose to conduct a population-based case-control study of renal cell cancer in areas of the U.S. with a high proportion of African American residents. We will include two study centers and one data coordinating center and will recruit study participants over a period of four years. We plan to conduct in-person interviews with 2,100 cases (1,400 whites and 700 blacks) and 2,800 controls (1,400 each of whites and blacks) to elicit information on demographic background and history of exposures. A 40 ml blood sample will be collected from living cases and controls to measure certain environmental exposures and for genetic analyses. Two buccal cell samples will be collected from living cases and controls for genetic analyses. Tumor tissue blocks will be collected from as many cases as possible for assays of tumor mutations. Diagnostic slides will be collected for standardized reclassification of tumors into clear cell, papillary, and other histologic subtypes. Medical records for all cases will be reviewed for health insurance coverage, concomitant conditions, presenting symptoms, tumor stage, size and grade, and methods leading to diagnosis of renal cell cancer.

DETAILED DESCRIPTION:
Incidence rates of renal cell cancer have increased rapidly in the U.S. and other countries. In particular, rates among African Americans have risen more sharply than any other cancer site. We propose to conduct a population-based case-control study of renal cell cancer two areas of the U.S. with a high proportion of African American residents: Detroit, Michigan (Wayne State University), and Chicago, Illinois (University of Illinois at Chicago). Westat, Inc. is the coordinating center. Participants are being recruited over a period of four years. A total of 2,100 cases (1,400 Caucasian Americans and 700 African Americans) and 2,800 controls (1,400 each of Caucasian and African Americans) will be recruited. In-person interviews are conducted with cases and controls to elicit information on demographic background and history of exposures. A 40 ml blood sample and a buccal cell sample are collected from cases and controls for genetic analyses. Tumor tissue blocks will be collected from as many cases as possible for assays of tumor mutations. Diagnostic slides will be collected for standardized reclassification of tumors into clear cell, papillary, and other histologic subtypes. Medical records for all cases will be reviewed for presenting symptoms, tumor stage, size and grade, and methods leading to diagnosis of renal cell cancer. Telephone interviews are conducted with the nest-of-kin of eligible cases who died before we could interview them. Permission is being sought from the next-of-kin to assess the case's medical records and obtain tumor tissue samples.

ELIGIBILITY:
* INCLUSION CRITERIA - CASES:

Residents of the study areas who are diagnosed with histologically confirmed renal cell carcinoma at ages 20 to 79 years over a four year study will be potentially eligible for the study.

In addition, only eligible patients who are mentally/physically able to provide informed consent and undergo interviews will be approached for participation.

INCLUSION CRITERIA - CONTROLS:

Population-based controls will be frequency-matched to the cases by study center, race, age and sex, at the ratio of one control per case for non-African Americans and two controls per case for African Americans.

Controls aged 65 years and older will be identified from Health Care Financing Administration (HCFA) files.

Controls under age 65 years will be identified from residents of the study areas by random telephone digit dialing (RDD).

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases and controls are residents of Chicago (Cook County), IL and Detroit (Wayne, Oakland, Macomb Counties), MI.
Sampling Method: Probability Sample
Enrollment: 2424 (Actual)
Dates: Start 2001-11-16 (Actual); Primary Completion 2007-01-31 (Actual); Study Completion 2016-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Purdue, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Wayne State University, Detroit, Michigan

REFERENCES:
- [Background] Bergstrom A, Moradi T, Lindblad P, Nyren O, Adami HO, Wolk A. Occupational physical activity and renal cell cancer: a nationwide cohort study in Sweden. Int J Cancer. 1999 Oct 8;83(2):186-91. doi: 10.1002/(sici)1097-0215(19991008)83:23.0.co;2-6. PMID 10471525
- [Background] Brauch H, Weirich G, Hornauer MA, Storkel S, Wohl T, Bruning T. Trichloroethylene exposure and specific somatic mutations in patients with renal cell carcinoma. J Natl Cancer Inst. 1999 May 19;91(10):854-61. doi: 10.1093/jnci/91.10.854. PMID 10340905
- [Background] Bruning T, Lammert M, Kempkes M, Thier R, Golka K, Bolt HM. Influence of polymorphisms of GSTM1 and GSTT1 for risk of renal cell cancer in workers with long-term high occupational exposure to trichloroethene. Arch Toxicol. 1997;71(9):596-9. doi: 10.1007/s002040050432. PMID 9285043